CLINICAL TRIAL: NCT02242318
Title: A Prospective, Randomised, Double-blind, Double-dummy Trial to Compare the Efficacy of Micardis® (Telmisartan) (80 mg p.o. Once Daily) and Valsartan (160 mg p.o. Once Daily) in Patients With Mild-to-moderate Hypertension After Missing One Dose Using Ambulatory Blood Pressure Monitoring
Brief Title: Study to Evaluate Efficacy of Micardis® (Telmisartan) and Valsartan in Patients With Mild-to-moderate Hypertension After Missing One Dose Using Ambulatory Blood Pressure Monitoring
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 502.376
Record Dates: First submitted 2014-09-16; First posted 2014-09-17 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan; Valsartan

ARMS (3):
- Telmisartan (Experimental): low dose for two weeks, then up titration to high dose, once daily
  Interventions: Drug: Telmisartan; Drug: Placebo
- Valsartan (Active Comparator): low dose for two weeks, then up titration to high dose, once daily
  Interventions: Drug: Valsartan; Drug: Placebo
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Telmisartan
  Arms: Telmisartan
Drug: Valsartan
  Arms: Valsartan
Drug: Placebo

SUMMARY:
The primary aim of the trial is to compare telmisartan 80 mg to valsartan 160 mg in lowering diastolic blood pressure in patients who missed a dose of their medication, as measured by ABPM (change from baseline in mean DBP over 24 hours), and to compare telmisartan 80 mg to valsartan 160 mg in lowering DBP during the last six hours of the dosing interval at the end of a 6 to 8-week treatment period, as measured by ABPM (change from baseline)

ELIGIBILITY:
Inclusion Criteria:

1. Mild-to-moderate hypertension defined as a mean seated diastolic blood pressure of ≥ 95 mmHg and ≤ 109 mmHg, measured by manual cuff sphygmomanometer, at Visit 2
2. 24-hour mean DBP of ≥ 85 mmHg at Visit 3 as measured by ABPM
3. Age 18 years or older
4. Ability to stop any current antihypertensive therapy without risk to the patient (investigator's discretion)
5. Patient's written informed consent in accordance with Good Clinical Practice (GCP) and local legislation

Exclusion Criteria:

1. Pre-menopausal women (last menstruation ≤ 1 year prior to start of run-in period) who

   1. are not surgically sterile,
   2. are nursing,
   3. are of child-bearing potential and are NOT practising acceptable methods of birth control, or do NOT plan to continue practising an acceptable method throughout the study. Acceptable methods of birth control include oral, implantable or injectable contraceptives and Intra Uterine Devices (IUD)
2. Known or suspected secondary hypertension
3. Mean sitting SBP ≥180 mmHg or mean sitting DBP ≥110 mmHg during any visit of the placebo run-in period
4. Hepatic and/or renal dysfunction as defined by the following laboratory parameters:

   1. Serum Glutamate-Pyruvate-Transaminase (Alanine Aminotransferase) (SGPT (ALT)) or Serum Glutamate-Oxaloacetate-Transaminase (Aspartate Aminotransferase) (SGOT (AST)) > than 2 times the upper limit of normal range,
   2. Serum creatinine > 2.3 mg/dL (or > 203 μmol/l)
5. Bilateral renal artery stenosis, renal artery stenosis in a solitary kidney, patients postrenal transplant or with only one kidney
6. Clinically relevant sodium depletion, hypokalaemia or hyperkalaemia
7. Uncorrected volume depletion
8. Primary aldosteronism
9. Hereditary fructose intolerance
10. Biliary obstructive disorders
11. Patients who have previously experienced symptoms characteristic of angioedema during treatment with ACE inhibitors or angiotensin II receptor antagonists
12. History of drug or alcohol dependency within six months prior to start of run-in period
13. Concomitant administration of any medications known to affect blood pressure, except medication allowed by the protocol
14. Any investigational therapy within one month of signing the informed consent form
15. Congestive heart failure (New York Heart Association (NYHA) functional class Congestive Heart Failure (CHF III-IV))
16. Unstable angina within the past three months prior to start of run-in period
17. Stroke within the past six months prior to start of run-in period
18. Myocardial infarction or cardiac surgery within the past three months prior to start of run-in period
19. Percutaneous Transluminal Coronary Angioplasty (PTCA) within the past three months prior to start of run-in period
20. Sustained ventricular tachycardia, atrial fibrillation, atrial flutter or other clinically relevant cardiac arrhythmias as determined by the investigator
21. Hypertrophic obstructive cardiomyopathy, aortic stenosis, hemodynamically relevant stenosis of the aortic or mitral valve
22. Patients with insulin-dependent diabetes mellitus whose diabetes has not been stable and controlled for at least the past three months as defined by an HbA1C ≥ 10%
23. Night shift workers who routinely sleep during the daytime and whose work hours include midnight to 4:00 Ante Meridiem (AM)
24. Known hypersensitivity to any component of the formulations
25. Any clinical condition which, in the opinion of the investigator would not allow safe completion of the protocol and safe administration of trial medication
26. Inability to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2001-09; Primary Completion 2002-09 (Actual)

PRIMARY OUTCOMES:
Change in 24 hour mean Diastolic blood pressure (DBP) after a missed dose | Baseline, Day 41, Day 55
  measured by ambulatory blood pressure monitoring (ABPM)
Change in mean DBP during the last 6 hours of the 24 hour dosing interval | up to 8 weeks

SECONDARY OUTCOMES:
Change in 24-hour mean systolic blood pressure (SBP) after a missed dose | Baseline, Day 41, Day 55
Change in mean SBP during the last 6 hours of the 24-hour dosing interval | up to 8 weeks
Change in pulse pressure (PP) | up to 8 weeks
Change in 24-hour mean DBP after an active dose of study medication | up to 8 weeks
Change in 24-hour mean SBP after an active dose of study medication | up to 8 weeks
Change in mean seated trough SBP/DBP/PP in- clinic manual cuff sphygmomanometer after a missed dose | up to 8 weeks
Change in the mean seated trough SBP/DBP/PP in- clinic manual cuff sphygmomanometer after an active dose of study medication | up to 8 weeks
Responder rate measured by ABPM after a missed dose of study medication | Baseline, Day 41, Day 55
  * ABPM DBP "control" (24-hour mean DBP < 80 mmHg),
  * ABPM DBP "response" (24-hour mean DBP < 80 mmHg and/or reduction from baseline ≥ 10 mmHg),
  * ABPM SBP "response" (24-hour mean SBP < 130 mmHg and/or reduction from baseline ≥ 10 mmHg)
Responder rate measured by ABPM after an active dose of study medication | up to 8 weeks
  * ABPM DBP "control" (24-hour mean DBP < 80 mmHg),
  * ABPM DBP "response" (24-hour mean DBP < 80 mmHg and/or reduction from baseline ≥ 10 mmHg),
  * ABPM SBP "response" (24-hour mean SBP < 130 mmHg and/or reduction from baseline ≥ 10 mmHg)
Responder rate in- clinic manual trough cuff measurements after a missed dose of study medication | Baseline, Day 41, Day 55
  * DBP "control" (DBP < 90 mmHg),
  * DBP "response" (DBP < 90 mmHg and/or fall of ≥ 10 mmHg),
  * SBP "response" (SBP < 140 mmHg and/or fall of ≥ 10 mmHg),
  * BP "normal" (SBP < 130 mmHg and DBP < 85 mmHg),
  * BP "normal / high normal" (SBP < 140 mmHg and DBP < 90 mmHg).
Responder rate in- clinic manual trough cuff measurements after an active dose of study medication | up to 8 weeks
  * DBP "control" (DBP < 90 mmHg),
  * DBP "response" (DBP < 90 mmHg and/or fall of ≥ 10 mmHg),
  * SBP "response" (SBP < 140 mmHg and/or fall of ≥ 10 mmHg),
  * BP "normal" (SBP < 130 mmHg and DBP < 85 mmHg),
  * BP "normal / high normal" (SBP < 140 mmHg and DBP < 90 mmHg).
Number of patients with adverse events | up to 8 weeks
Change in 24-hour Pulse Pressure (PP) after a missed dose | Baseline, Day 41, Day 55